CLINICAL TRIAL: NCT06921564
Title: Effects of Lower-body Strength Training Combined With Small-sided Games on Physical Performance in Young Soccer Players
Brief Title: Effects of Combined Training on Physical Performance in Young Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Muhammet Taha İlhan, Research Assistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AdnanMU-FSS-MTI-577954-280325-
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Young Soccer Players
Keywords: Small-sided games; strength training; combined training; physical performance; soccer

STUDY DESIGN:
Intervention Model Description: This study used a randomized matched-pairs design. The players were ranked according to their Yo-Yo Intermittent Recovery Test Level 1 results and then paired on the basis of these rankings. On the basis of these data, they were then randomly assigned to one of two groups: (1) CT (strength training + small-sided games) and (2) Small-sided games alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Training (Experimental): During the 6-week intervention period, the combined training group performed 2 sessions per week of lower-body strength training and 2 sessions per week of small-sided games training in different formats. The combined training group also participated in their team's regular soccer training, which focused on technical and tactical skills, with 5 sessions per week (60-90 minutes each).
  Interventions: Other: Combined training
- Small-sided games alone (Experimental): The small-sided games group performed 2 sessions per week of small-sided games training program in different formats, without participating in any strength training. The combined training group also participated in their team's regular soccer training, which focused on technical and tactical skills, with 5 sessions per week (60-90 minutes each).
  Interventions: Other: Small-sided games alone

INTERVENTIONS:
Other: Combined training — During the 6-week intervention period, the combined training group performed 2 sessions per week of lower-body strength training and 2 sessions per week of small-sided games training in different formats. The strength training was performed on Tuesdays and Thursdays. This training was finished at least one hour before the team's technical and tactical soccer training. The strength training program is designed to include movements for bilateral hip dominant, bilateral knee dominant, unilateral hip dominant, unilateral knee dominant and calf muscles. The exercises were selected to allow players to perform them on the field with minimal equipment, without the need for machines. In addition, small field games training was practiced two days a week. Repetitions in reserve and resistance training-specific ratings of the perceived exertion scale were used to determine training intensity and load.
  Arms: Combined Training
Other: Small-sided games alone — The small-sided games group performed 2 sessions per week of small-sided games training program in different formats, without participating in any strength training. The small-sided games training was conducted twice a week on Wednesdays and Fridays (8:00-10:00 p.m.) for 6 weeks. These training sessions started before the team's technical and tactical training. Extra balls are placed at the goals and along the field boundary lines, allowing play to restart immediately after the ball leaves the field. During the games, the offside rule was not applied. The game started with the foot when the ball left edge of the field. Other rules in the games were kept similar to those of official soccer. During the games, the coaches encouraged the players to exert maximum effort. The number of defenders, midfielders, and attackers in the teams was kept as equal as possible.
  Arms: Small-sided games alone

SUMMARY:
Small-sided games (SSGs) are an effective training method for improving aerobic fitness. However, their effects on physical performance attributes such as, sprinting, jumping, agility, and repeated sprint ability (RSA) remain unclear. Therefore, this study aimed to compare the effects of lower-body strength training combined with SSGs training (CT) versus SSGs training alone on sprinting, agility, RSA, countermovement jump (CMJ), and aerobic fitness in young soccer players. Twenty young soccer players were randomly assigned to one of two groups: CT (n = 10; age: 14.0 ± 0.0) and SSGs (n = 10; age: 14.0 ± 0.0). The CT group performed lower-body strength training twice a week, in addition to SSGs training twice a week. The SSGs group performed SSGs training only twice a week, without any strength training. Before and after the 6-week training intervention, the 20-m sprint test, Illinois agility test (IAT), RSA, CMJ, and Yo-Yo Intermittent Recovery Test Level 1 were conducted.

ELIGIBILITY:
Inclusion Criteria:

* have no injuries, illnesses, or physical limitations that would prevent participation in the study
* have been training and playing official soccer for a minimum of 2 years
* have participated in all testing protocols
* have participated in a minimum of 80% of the training sessions
* have not participated in any structured strength training program for the last six months, except for bodyweight exercises; and
* have not been a goalkeeper

Ages: 14 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Height | After 6 weeks of training intervention
  Height (in cm) was measured using a stadiometer (SECA, Hamburg, Germany). These measurement was taken in the morning, before breakfast, while the players wore light clothing and no shoes. Measurement was performed twice to reduce the margin of error.
Body weights | After 6 weeks of training intervention
  Body weights (in kg) were measured using a body mass measuring device (Fakir, Germany). These measurement was taken in the morning, before breakfast, while the players wore light clothing and no shoes. Measurement was performed twice to reduce the margin of error.
Body mass index | After 6 weeks of training intervention
  Body mass index (BMI) (kilograms/m2) was calculated from height and body weight values.
20-m sprint | After 6 weeks of training intervention
  The sprinting performance was assessed using the 20-m linear sprint test. The test was conducted using two pairs of photocells (Smartspeed, Fusion Sport Pty Queensland, Australia). The starting point was placed 70 cm behind the first pair of photocells. First, a familiarization trial was conducted at low intensity. The test was then performed twice, with two-minute passive recovery intervals. The best result was used for analysis.
Agility | After 6 weeks of training intervention
  To assess agility performance, the Illinois Agility Test (IAT), a valid and reliable test for male team athletes, was used. Prior to starting the test, the player lies in a prone position, with the chin touching the surface of the starting line. After the researcher's command started, the player quickly stood up and ran in the indicated direction, avoiding contact with the placed cones. First, a familiarization trial was conducted at low intensity. Two trials were then performed, with two-minute passive recovery intervals. The best time was used for analysis.
Repeated sprint ability (RSA) | After 6 weeks of training intervention
  RSA was assessed using the 6x20-m RSA test. A 20-second rest interval was provided between sprints. A photocell system (Smartspeed, Fusion Sport Pty, Queensland, Australia) was placed at the start and at the 20-m line to measure sprint time. The players started the test from the line marked 70 cm behind the first pair of photocells. The mean sprint time (mean sprint time over the six sprints) (RSAmean) and the total sprint time (total time over the six sprints) (RSAtotal) were used for the analysis.
Vertical jump | After 6 weeks of training intervention
  Vertical jump performance was evaluated using the countermovement jump (CMJ) test. The test was performed using the My Jump Lab smartphone application (Spain, Madrid, version 1.2.2), which has proven validity and reliability for vertical jump measurement. Players were instructed to begin the jump with their feet shoulder-width apart, in a 90° knee flexion position, with their hands on their hips. During the test, players were instructed to jump as high as possible while keeping their hands on their hips. The mobile phone was positioned 3 meters away from the player, and the camera height was set to 0.90 meters using a tripod. The players first performed a familiarization trial at low intensity. Each player then performed three jumps, with two-minute passive recovery intervals. The highest jump was used for analysis
Aerobic fitness | After 6 weeks of training intervention
  Aerobic fitness was assessed using the Yo-Yo Intermittent Recovery Test Level 1 (YYIRTL-1). The test was conducted following previously described instructions (Bangsbo et al., 2008). The players' estimated maximum oxygen consumption (VO2max) after the test was calculated using the formula ''VO2max = 36.4 + (0.0084 x covered distance in YYIRTL-1)''.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want to make any statement.

REFERENCES:
- [Background] Querido SM, Clemente FM. Analyzing the effects of combined small-sided games and strength and power training on the fitness status of under-19 elite football players. J Sports Med Phys Fitness. 2020 Jan;60(1):1-10. doi: 10.23736/S0022-4707.19.09818-9. PMID 32008309
- [Background] Arslan E, Soylu Y, Clemente FM, Hazir T, Kin Isler A, Kilit B. Short-term effects of on-field combined core strength and small-sided games training on physical performance in young soccer players. Biol Sport. 2021 Oct;38(4):609-616. doi: 10.5114/biolsport.2021.102865. Epub 2021 Feb 11. PMID 34937971